CLINICAL TRIAL: NCT00288717
Title: A Randomized, Comparative Study of the Effects of Candesartan and Telmisartan on the Home Blood Pressure, Glucose and Lipid Metabolism in the Hypertensive Patients With the Accumulation of Visceral Fat by the Central Registration System
Brief Title: Effectiveness of Candesartan and Telmisartan on Morning Hypertension in Japanese Obese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saitama Medical University (Other)
Collaborators: Non-Profit Organaizaion "LINE" (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUJIYAMA-Study; UMIN-CTR-C000000324
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2007-01-11 (Estimated); Status verified 2007-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan; Telmisartan

INTERVENTIONS:
Drug: Candesartan
Drug: Telmisartan

SUMMARY:
To investigate the effects of Candesartan and Telmisartan on the home blood pressure, glucose and lipid-metabolism in the hypertensive patients with the accumulation of visceral fat by the newly developed Tele-medicine system

DETAILED DESCRIPTION:
A randomized, comparative study of the effects of Candesartan and Telmisartan on the home blood pressure, glucose and lipid metabolism in the hypertensive patients with the accumulation of visceral fat by the central registration system

ELIGIBILITY:
Inclusion Criteria:

* Circumference at waist: male ≧85 cm, female ≧90 cm
* Hypertensive patient with untreated hypertension, and casual blood pressure of systole ≧140 mmHg, or diastole ≧90 mmHg
* Hypertensive patient with hypertension under treatment, and casual blood pressure of systole ≧130 mmHg, or diastole ≧85 mmHg

Exclusion Criteria:

* Significant hypertensive patient with diastolic blood pressure ≧120 mmHg
* Malignant hypertensive patient
* Patient with a contraindication to the study drugs (hypersensitivity, significant hepatic diseases, pregnant woman)
* Patient with urinary protein (qualitative) ＋～＋＋
* Patient with familial hyperlipidemia
* Other patients judged as ineligible for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2006-02; Study Completion 2007-09

PRIMARY OUTCOMES:
Home blood pressure in the early morning

SECONDARY OUTCOMES:
Home blood pressure at bedtime
M/E ratio
Casual blood pressure
Body fat percentage
Body weight
Height
BMI
Blood potassium
Total cholesterol
HDL cholesterol
LDL cholesterol
Triglyceride
Blood glucose
IRI
HbAlc*
HOMA-IR
Urinary trace albumin
Creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Hidetomo Nakamoto, MD, Principal Investigator — Saitama Medical School Department of Renal Medicine
Locations (1):
- Saitama Medical School Department of Renal Medicine, Saitama, Saitama, Japan